CLINICAL TRIAL: NCT04508296
Title: De-escalation Fluid Management Guided by Volumetric Parameters in Patients With Sepsis and ARDS
Brief Title: The Effect pf Goal-directed De-escalation in ARDS on Organ Function and Mortality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern State Medical University (Other)
Responsible Party: Principal Investigator, Mikhail Y. Kirov, Head of Department, Northern State Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: De-escalation ARDS_2016
Record Dates: First submitted 2020-08-05; First posted 2020-08-11 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: ARDS, Human; Sepsis, Severe
Keywords: de-escalation therapy; acute respiratory distress syndrome; extravascular lung water; global end-diastolic volume; sepsis
MeSH Terms: conditions — Respiratory Distress Syndrome; Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GEDVI-oriented de-escalation (Experimental): Patients received de-escalation fluid management using either diuretics or ultrafiltration during continuous RRT. In the case of GEDVI > 650 mL/m2 the primary goal of de-escalation is to obtain a cumulative fluid balance after 48 hrs from the study baseline of 0 to -3000 mL. In the case of GEDVI < 650 mL/m2 he target fluid balance is in the range of 0 to +3000 mL
  Interventions: Diagnostic Test: Goal directed de-escalation therapy
- EVLWI-oriented de-escalation (Experimental): Patients received de-escalation fluid management using either diuretics or ultrafiltration during continuous RRT. In the case of EVLWI > 10 mL/kg the primary goal of de-escalation is to obtain a cumulative fluid balance after 48 hrs from the study baseline of 0 to -3000 mL. In the case of EVLWI < 10 mL/kg, the target fluid balance is in the range of 0 to +3000 mL
  Interventions: Diagnostic Test: Goal directed de-escalation therapy

INTERVENTIONS:
Diagnostic Test: Goal directed de-escalation therapy — Patients received de-escalation fluid management using either diuretics or ultrafiltration during continuous RRT in the case of GEDVI > 650 mL/m2 or EVLWI > 10 mL/kg depending on the randomization group. The primary goal of de-escalation was to obtain a cumulative fluid balance after 48 hrs from the study baseline of 0 to -3000 mL. In the case of GEDVI < 650 mL/m2 or EVLWI < 10 mL/kg, the target fluid balance was in the range of 0 to +3000 mL

SUMMARY:
Objective: To compare two de-escalation strategies guided by either extravascular lung water or global end-diastolic volume-oriented algorithms in patients with sepsis and ARDS.

Design: A prospective randomized study. Setting: City Hospital #1 of Arkhangelsk, Russia, mixed ICU. Patients: Sixty patients with sepsis and ARDS were randomized to receive de-escalation fluid therapy, guided either by extravascular lung water index (EVLWI, n = 30) or global end-diastolic volume index (GEDVI, n = 30).

Intervention: In case of GEDVI > 650 mL/m2 or EVLWI > 10 mL/kg, diuretics and/or controlled ultrafiltration were administered. The primary goal of de-escalation was to achieve the cumulative 48-hr fluid balance in the range of 0 to - 3000 mL. If GEDVI < 650 mL/m2 or EVLWI < 10 mL/kg, the target fluid balance was set from 0 to +3000 mL.

DETAILED DESCRIPTION:
In all patients, investigators catheterized the internal jugular or the subclavian vein with a triple-lumen central venous catheter (Certofix, B|Braun, Germany) and the femoral artery with a thermistor-tipped arterial catheter (5F, PV2015L20, Pulsion Medical Systems, Munich, Germany). The arterial blood pressure was recorded from a side port of the catheter. Hemodynamic monitoring was carried out using the method of transpulmonary thermodilution (PiCCO2 monitor, Pulsion Medical Systems, Germany) by a triplicate 15 mL bolus of cold (< 8 °C) 0.9% saline solution.

Mechanical ventilation (Puritan Bennett 840 and 980, Medtronic, USA) was performed according to the ARDS Network protocol, using pressure-controlled ventilation with tidal volume 6-7 ml/kg of predicted body weight, with a Ppeak not exceeding 35 cm H2O, positive end-expiratory pressure (PEEP) and a fraction of inspiratory oxygen (FiO2) levels adjusted to maintain SpO2 within a 92-97% range.

The target fluid balance was achieved by continuous infusion of furosemide with an initial dose of 0.07 mcg/kg/hr and a minimal duration of 12 hrs. In case of failure to reach a negative fluid balance by means of diuretics, started controlled ultrafiltration using continuous veno-venous hemofiltration (CVVH, multiFiltrate, Fresenius Medical Care, Germany). For fluid replacement, if necessary, investigators administered balanced crystalloid solutions (Sterofundin Iso/G5, B|Braun, Germany) with an initial infusion rate of 6-7 ml/kg/hr.

Heart rate (HR), MAP, cardiac index (CI), GEDVI, EVLWI, pulmonary vascular permeability index (PVPI), central venous pressure (CVP), systemic vascular resistance index (SVRI), pulse pressure variation (PPV), and stroke volume variation (SVV) were assessed using transpulmonary thermodilution and arterial pulse contour analysis. During the study, investigators also assessed blood gases (ABL Flex 800 Radiometer, Denmark) and biochemical parameters (Random Access A-25, BioSystems, Spain). All measurements were performed at baseline, at 24 and at 48 hrs of the goal-directed de-escalation

ELIGIBILITY:
Inclusion Criteria:

* The presence of sepsis ( the third international definition of sepsis and septic shock )
* The precence of ARDS (the Berlin definition of ARDS)
* mechanical ventilation before the study for at least 24 hrs
* the age of the patient > 18 years.

Exclusion Criteria:

* continuous infusion of norepinephrine in a dose exceeding 0.4 mcg/kg/min to maintain mean arterial pressure (MAP) within 65-75 mm Hg,
* morbid obesity with BMI > 40 kg/m2,
* severe brain injury,
* chronic kidney diseases,
* pregnancy,
* known irreversible underlying conditions such as end-stage neoplasms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-03-10 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
Improvement of organ function | 48 hours
  To assess if ELWI- or GEDVI-oriented goal-directed therapy can lead to the decrement of the SOFA scale by more than 20% in comparison with baseline values.

SECONDARY OUTCOMES:
Survival | 28-day
  The secondary endpoint was to evaluate whether ELWI- or GEDVI-oriented goal-directed therapy can lead to the decrement of the 28-days mortality

CONTACTS AND LOCATIONS:
Locations (1):
- City Hospital # 1 n.a. E.E. Volosevich, Arkhangelsk, Russia

IPD SHARING:
Plan to Share IPD: Undecided